CLINICAL TRIAL: NCT06786806
Title: The Impact of Gamified Infection Control Education on Academic Self-Efficacy, Learning Motivation, and Cognitive Achievement in Nursing Students: A Randomized Controlled Trial
Brief Title: Gamified Infection Control Education for Nursing Students: Effects on Self-Efficacy, Motivation, and Learning Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Beratiye Oner, Assistant Professor, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024071
Record Dates: First submitted 2025-01-11; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Students, Nursing
Keywords: Gamification; infection control; nursing student; academic success; self efficacy

STUDY DESIGN:
Intervention Model Description: This study utilized a randomized controlled trial (RCT) design, where participants were randomly assigned to one of two groups. The intervention group (n=30) participated in a four-week Gamified Infection Control Education Program that included interactive components such as physical games, case studies, and escape rooms. In contrast, the control group (n=30) received traditional lecture-based instruction, serving as the comparator. This design aimed to evaluate the effectiveness of gamification in enhancing student engagement, motivation, and learning outcomes compared to standard educational methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who received the Gamified Infection Control Education Program.
  Interventions: Other: Gamified Infection Control Education Program
- Control (Other): Participants who received traditional lecture-based instruction.
  Interventions: Other: Traditional Lecture-Based Instruction

INTERVENTIONS:
Other: Gamified Infection Control Education Program — A four-week educational program integrating gamification techniques such as physical games, case studies, and escape rooms to teach infection control practices.Designed to enhance engagement, learning motivation, and cognitive achievement among nursing students.
  Arms: Intervention
Other: Traditional Lecture-Based Instruction — Standard didactic teaching method focusing on infection control principles without incorporating gamification. Served as the comparator to evaluate the effectiveness of the gamified program.
  Arms: Control

SUMMARY:
Infection control is a critical component of nursing education, ensuring the safety of patients and healthcare workers. Gamification, which integrates game-based principles into educational activities, has emerged as a promising approach to improve student engagement, motivation, and learning outcomes in healthcare education. This study aimed to evaluate the impact of a gamified infection control education program on cognitive achievement, academic self-efficacy, and learning motivation among first-year nursing students. The study employed a randomized controlled trial design involving 60 first-year nursing students from a private university in Turkey. Participants were randomly assigned to an intervention group (n=30) or a control group (n=30). The intervention group participated in a four-week Gamified Infection Control Program featuring physical games, case studies, and escape rooms. The control group received traditional lecture-based instruction. Data were collected using validated instruments, including the Infection Control Cognitive Achievement Measurement Questions Form, the Academic Nurse Self-Efficacy Scale (ANSES), and the Learning Motivation Scale in Higher Education (EMAPRE-U). Statistical analyses included t-tests, Mann-Whitney U tests, and regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing students enrolled in a nursing program
* Students who have not previously completed formal infection control training
* Students who are willing to participate in the study and provide informed consent

Exclusion Criteria:

* Students with prior knowledge or certification in infection control practices
* Students who are unable to attend the full four-week program due to scheduling conflicts
* Students with any medical or psychological condition that would prevent full participation in study activities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Cognitive Achievement in Infection Control | Assessed immediately after the four-week intervention.
  Improve cognitive understanding of infection control principles, including sterilization and sepsis practices. The investigators used the Infection Control Cognitive Achievement Measurement Questions Form as the measurement tool. Each question has a single correct answer. Each correct answer is worth one point, and higher total scores reflect higher levels of The Infection Control Cognitive Achievement Measurement. The lowest total score is '0' and the highest total score is '100'.

SECONDARY OUTCOMES:
Learning Motivation | Assessed immediately after the four-week intervention.
  Change in learning motivation levels among nursing students. The investigators used the Learning Motivation Scale in Higher Education as the measurement tool. Participants select their level of agreement about (item) using a Likert scale ranging from 1 (disagree) to 3 (agree). Higher scores reflect higher motivation to learn. The lowest total score is '23' and the highest total score is '69'.
Academic Self-Efficacy | Assessed immediately after the four-week intervention.
  Change in students' confidence in their academic abilities related to infection control. The investigator used the Academic Nurse Self-Efficacy Scale as the measurement tool. Participants respond to the prompt, "How confident are you about (item)?" using a Likert scale ranging from 1 (very little confidence) to 5 (completely confident). Higher scores reflect greater levels of academic self-efficacy. The lowest total score is '14' and the highest total score is '70'.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No